CLINICAL TRIAL: NCT01976195
Title: An Open-label, Randomized Multicenter Investigation of High-dose Dexamethasone Combining Thalidomide Versus High-dose Dexamethasone Mono-therapy for Management of Newly-diagnosed Immune Thrombocytopenia
Brief Title: High-dose Dexamethasone Combining Thalidomide Versus Dexamethasone Mono-therapy for Management of Newly-diagnosed ITP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Collaborators: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other); Anhui Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Thalidomide
Record Dates: First submitted 2013-10-21; First posted 2013-11-05 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2013-10

CONDITIONS: Immune Thrombocytopenia
Keywords: Thalidomide; Dexamethasone; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide plus HD-Dexmamethasone (Experimental): Thalidomide 150mg per day, 15 consecutive days Dexamethasone 40 mg per day, 4 consecutive days
  Interventions: Drug: Dexamethasone; Drug: Thalidomide
- Dexamethasone (Active Comparator): Dexamethasone 40 mg per day, 4 consecutive days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 40 mg per day, 4 consecutive days
Drug: Thalidomide — Thalidomide 150mg per day, 15 consecutive days
  Arms: Thalidomide plus HD-Dexmamethasone

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of thalidomide combining with high-dose dexamethasone for the treatment of adults with primary immune thrombocytopenia (ITP), compared to conventional high-dose dexamethasone mono-therapy.

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter, randomized controlled trial of 200 primary ITP adult patients from 5 medical centers in China. One part of the participants are randomly selected to receive Thalidomide (given at a dose of 150mg for 15 consecutive days), combining with dexamethasone (given intravenously at a dose of 40 mg per day for 4 days, the others are selected to receive high-dose of dexamethasone treatment (given intravenously at a dose of 40 mg daily for 4 days).

Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of thalidomide combining with high-dose dexamethasone therapy compared to high-dose dexamethasone for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

* •newly diagnosed ITP patients need of treatment(s) to minimize the risk of clinically significant bleeding primary ITP confirmed by excluding other supervened causes of thrombocytopenia

Exclusion Criteria:

* •pregnancy hypertension cardiovascular disease diabetes liver and kidney function impairment hepatitis C virus, HIV, HBsAg seropositive status patients with systemic lupus erythematosus and/or antiphospholipid syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response | Newly diagnosed ITP in 3 months
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China